CLINICAL TRIAL: NCT02429713
Title: The Effects of Tourniquet Use in Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: The Effects of Tourniquet Use in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Wang Kai, resident, Peking University People's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PekingUPH
Record Dates: First submitted 2015-04-15; First posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Blood Loss
Keywords: tourniquet; total knee arthroplasty; blood loss
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short-duration tourniquet group (Experimental): The tourniquet was inflated immediately before cement application and deflated after its hardening
  Interventions: Procedure: Short-duration tourniquet
- Long-duration tourniquet group (Active Comparator): The tourniquet was inflated immediately before incision and deflated after the hardening of the cement
  Interventions: Procedure: Long-duration tourniquet

INTERVENTIONS:
Procedure: Short-duration tourniquet — Short-duration tourniquet group:inflate the tourniquet immediately before cement application and deflated after its hardening
  Arms: Short-duration tourniquet group
Procedure: Long-duration tourniquet — Long-duration tourniquet group: inflate the tourniquet immediately before incision and deflated after the hardening of the cement
  Arms: Long-duration tourniquet group

SUMMARY:
Tourniquets are still widely used in total knee arthroplasty, but are associated with several adverse effects. Most of previous studies did not randomize the participants so the baseline difference of the patients might have influenced the outcome. Therefore, investigators conducted a randomized controlled trial, in which all the patients received staged bilateral TKA with two different durations of tourniquet use. Investigators aimed to quantify the effect of tourniquet use on reducing blood loss and to evaluate the impact of tourniquet use on functional and clinical outcome.

DETAILED DESCRIPTION:
Fifty participants who underwent staged bilateral TKA were recruited in this study. On one side, the tourniquet was inflated immediately before incision and deflated after the hardening of the cement. On the other side the tourniquet was inflated immediately before cement application and deflated after its hardening. Blood loss, operating time, transfusion rate, postoperative pain, limb swelling, deep vein thrombosis (DVT) incidence and clinical outcomes were monitored for comparison.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 50 years or over
* classified as American Society of Anesthesiologists ASA 1-2.

Exclusion Criteria:

* coagulopathy,
* uncontrolled hypertension,
* peripheral vascular disease and
* patients with BMI≥35

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | within operation

SECONDARY OUTCOMES:
Thigh pain measured by Visual Analogue Scale/Score (VAS) | 1 day, 2 day, 1 week, 2 week and 6 week after surgery
Thigh swelling measured by circumference 10 cm proximal to the patella | 1 day, 2 day, 1week, 2 week and 6 week after surgery
Postoperative blood loss measured by drainage volume | 1 day and 2 day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jianhao Lin, M.D., Study Director — Peking University People's Hospital

REFERENCES:
- [Background] Tai TW, Lin CJ, Jou IM, Chang CW, Lai KA, Yang CY. Tourniquet use in total knee arthroplasty: a meta-analysis. Knee Surg Sports Traumatol Arthrosc. 2011 Jul;19(7):1121-30. doi: 10.1007/s00167-010-1342-7. Epub 2010 Dec 15. PMID 21161177
- [Background] Hernandez AJ, Almeida AM, Favaro E, Sguizzato GT. The influence of tourniquet use and operative time on the incidence of deep vein thrombosis in total knee arthroplasty. Clinics (Sao Paulo). 2012 Sep;67(9):1053-7. doi: 10.6061/clinics/2012(09)12. PMID 23018303